CLINICAL TRIAL: NCT00295763
Title: Follow-up of Thyroid Cancer Patients From Study THYR-008-00 Who Received Thyroid Remnant Ablation Using Either the Hypothyroid or the Thyrogen Method.
Brief Title: A New Study to Follow-up Thyroid Cancer Patients Who Participated in a Previous Study, Which Compared the Success of Destruction of the Thyroid Remnant Using Standard Treatment or Thyrogen.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THYR01605
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Differentiated Thyroid Cancer
Keywords: papillary thyroid cancer; follicular thyroid cancer; recombinant human TSH; Thyrogen; thyroid stimulating hormone; thyroid remnant ablation; radioiodine
MeSH Terms: conditions — Thyroid Cancer, Papillary; Adenocarcinoma, Follicular | interventions — Thyrotropin Alfa; Injections

ARMS (1):
- 1 (Other)
  Interventions: Drug: Thyrogen (thyrotropin alfa for injection)

INTERVENTIONS:
Drug: Thyrogen (thyrotropin alfa for injection) — No reference therapy was given. All patients in this follow-up study received Thyrogen. Thyrogen 0.9 mg was administered intramuscularly (IM) in the buttock on 2 consecutive days.
  For WBS and static neck imaging, each patient received 4 mCi (148 MBq) ± 0.4 mCi 131I PO.

SUMMARY:
Patients diagnosed with thyroid cancer are commonly treated with surgery to remove their thyroid gland followed by radioiodine ablation to destroy any remaining parts of the thyroid gland that may have been missed during surgery. It is thought that ablation with radioiodine destroys normal remaining thyroid tissue as well as cancerous cells either in the thyroid area or at other sites.

Following successful treatment, patients are then monitored by their physicians at regular intervals with testing to detect any recurrence of thyroid cancer throughout the body. If thyroid cells are detected by these follow up tests, the physician will decide the best method to re-treat the patient.

In 2001-2003 Genzyme conducted a clinical study to test if Thyrogen® can be used to accomplish radioiodine ablation treatment. This study aimed to determine that the success rates of radioiodine ablation were comparable when patients were prepared for ablation with Thyrogen® while being maintained on their normal thyroid hormone therapy, or, alternatively, by thyroid hormone withdrawal. Thyroid hormone withdrawal commonly causes uncomfortable side effects for patients, and these might be avoided by the use of Thyrogen.

Eight months after the initial Thyrogen plus radioiodine treatment to achieve ablation, all patients in both groups were given Thyrogen® to test for any remaining thyroid tissue. The results of this testing showed that all patients (in both groups) had successfully achieved remnant ablation and had no detectable thyroid tissue remaining.

In order to confirm these remnant ablation results we will conduct follow up testing in this study for all patients that were enrolled in the previous study and we also will determine if their thyroid cancer has recurred. Only patients who completed this previous Thyrogen ablation study are eligible for entry into this study.

ELIGIBILITY:
Inclusion Criteria:

* Committed to follow the protocol requirements, as evidenced by providing written informed consent before any study-related procedures are performed and within 28 days prior to Day 1;
* Completed the THYR-008-00 study;
* A negative serum pregnancy test within 8 days prior to the start of the week during which the patient will receive Thyrogen and radioiodine (required for all pre-menopausal women of child bearing potential, with menopause defined as age >50 years with >2 years without a menstrual period)

Exclusion Criteria:

* Patients who are currently taking amiodarone or other prescribed iodine-containing medication;
* Patients who received iodine-containing X-ray contrast material within the prior 3 months;
* Women of child-bearing potential, unless confirmed to have a negative pregnancy test prior to dosing;
* Women who are pregnant or lactating;
* Patients who are currently participating in another investigational drug study or who have participated in such a study within 30 days of their enrollment in this study;
* Patients with schedule or travel plans that prevent the completion of all required visits;
* The patient who by mistake received only one-half the intended dose of Thyrogen during THYR-008-00 (Patient 209);
* The patient in THYR-008-00 who was found to have lung metastases on her post therapy scan (Patient 204);
* A concurrent major medical disorder (e.g., documented significant cardiac disease, debilitating cardiopulmonary disease, advanced renal failure, advanced liver disease, advanced pulmonary disease, or advanced cerebral vascular disorder) that may have an impact on the capability of the patient to adequately comply with the requirements of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To confirm the status of thyroid remnant ablation by using Thyrogen stimulated radioiodine whole body scans (WBS) in patients previously treated in THYR-008-00. | Duration of study
To learn if there was recurrence of thyroid cancer in any of the patients previously treated in the THYR-008-00 study. | Duration of study
To assess Thyrogen-stimulated serum Tg measurements in patients previously treated in the THYR-008-00 study. | Duration of study
To assess safety information on repeat exposure to Thyrogen in patients previously treated in the THYR-008-00 study. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (9):
- United States (4):
  - University of Colorado Health Sciences Centre, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Ohio State University, Columbus, Ohio
  - MD Anderson Cancer Centre, Houston, Texas
- LHRI Research Services, London, Ontario, Canada
- France (2):
  - Centre Rene Huguenin, Saint-Cloud
  - Institut Gustave Roussy, Villejuif
- University of Wurzburg, Würzburg, Germany
- University of Pisa, Pisa, Italy

REFERENCES:
- [Derived] Elisei R, Schlumberger M, Driedger A, Reiners C, Kloos RT, Sherman SI, Haugen B, Corone C, Molinaro E, Grasso L, Leboulleux S, Rachinsky I, Luster M, Lassmann M, Busaidy NL, Wahl RL, Pacini F, Cho SY, Magner J, Pinchera A, Ladenson PW. Follow-up of low-risk differentiated thyroid cancer patients who underwent radioiodine ablation of postsurgical thyroid remnants after either recombinant human thyrotropin or thyroid hormone withdrawal. J Clin Endocrinol Metab. 2009 Nov;94(11):4171-9. doi: 10.1210/jc.2009-0869. Epub 2009 Oct 22. PMID 19850694